CLINICAL TRIAL: NCT04871308
Title: Cardioprotective Effect of Dexmedetomidine in Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass: a Randomized, Placebo-controlled Trial
Brief Title: Dexmedetomidine and Myocardial Protection
Acronym: DEXCARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Karam Nam, MD, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEXCARD
Record Dates: First submitted 2021-05-03; First posted 2021-05-04 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Placebo Comparator): Placebo group using normal saline infusion
  Interventions: Drug: Control
- Dexmedetomidine (Active Comparator): From anesthesia induction before the initiation of cardiopulmonary bypass, dexmedetomidine is infused intravenously at a rate of 0.5 mcg/kg/hr after a loading dose infusion of 0.75 mcg/kg for 10 mins.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Anesthesia is induced using midazolam or etomidate, and sufentanil. A target-controlled infusion of propofol and remifentanil is used for anesthesia maintenance.
  From anesthesia induction before the initiation of cardiopulmonary bypass, dexmedetomidine is infused intravenously at a rate of 0.5 mcg/kg/hr after a loading dose infusion of 0.75 mcg/kg for 10 mins.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Control — During the same time window for dexmedetomidine, normal saline is infused at the same rate calculated for dexmedetomidine.
  Arms: Control

SUMMARY:
Dexmedetomidine, an alpha-2 agonist, is a sedative that is widely used in various clinical settings because, compared to benzodiazepines, it preserves respiratory function better and its duration of action is short.

Recent experimental studies showed a possibility that dexmedetomidine may have an organoprotective effect from ischemic-reperfusion injury by reducing inflammatory response. Besides, dexmedetomidine is known to be related with attenuated sympathetic tone and improved microcirculation.

Taken together, it is plausible that dexmedetomidine exerts cardioprotection in patients undergoing cardiac surgery with cardiopulmonary bypass and aortic cross-clamp.

The aim of this trial is to test the effect of dexmedetomidine on postoperative cardiac troponin I measurements in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgery utilizing cardiopulmonary bypass and aortic cross-clamp

Exclusion Criteria:

* Coronary artery bypass grafting
* Concomitant cryo-Maze procedure
* Myectomy
* Heart transplantation
* Concomitant major non-cardiac surgery
* Isolated complicated congenital heart surgery
* descending thoracic aorta surgery with partial cardiopulmonary bypass
* Emergency surgery
* Minimally invasive or robot-assisted surgery
* Estimated GFR <30 ml/min/1.73 m2
* Documented end-stage renal disease
* Preoperative renal replacement therapy
* Preoperative history of percutaneous coronary intervention within 6 month before surgery
* Acute coronary syndrome within 4 weeks before surgery
* Preoperative mechanical circulatory support devices

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
cardiac troponin I | Three days after surgery
  Area under the curve of cardiac troponin I measured at 0, 6, 24, 48, 72 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Karam Nam, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea